CLINICAL TRIAL: NCT03743298
Title: Phase 1B Trial of AV-MEL-1 (Autologous Dendritic Cells Loaded With Autologous Tumor Antigens) With Anti-PD-1 Checkpoint Inhibitors in Metastatic Melanoma
Brief Title: Safety of AV-MEL-1 With Anti-PD-1 Therapy in Metastatic Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aivita Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-MEL-P01-US
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AV-MEL-1 (Experimental): AV-MEL-1: Autologous dendritic cells loaded with autologous tumor antigens (ATA) from a short-term cell culture of autologous tumor cells. AV-MEL-1 is admixed with granulocyte-macrophage colony stimulating factor (GM-CSF) as an adjuvant, prior to injection.
  Interventions: Drug: AV-MEL-1

INTERVENTIONS:
Drug: AV-MEL-1 — AV-MEL-1: Autologous dendritic cells loaded with autologous tumor antigens (ATA) from a short-term cell culture of autologous tumor cells. AV-MEL-1 is admixed with granulocyte-macrophage colony stimulating factor (GM-CSF) as an adjuvant, prior to injection.

SUMMARY:
This is an open label, single-arm, phase IB treatment study to determine the safety of administering anti-PD1 monoclonal antibodies with AV-MEL-1 and to get some suggestion of efficacy, in patients with measurable metastatic melanoma. The study is open to patients who have either never received treatment for metastatic melanoma or were previously treated with anti-PD-1 with or without anti-CTLA-4 or with enzymatic inhibitors of the BRAF/MEK pathway because of BRAF600E/K mutations, and are about to initiate anti-PD-1 monotherapy. The intent is to treat 14 to 20 patients with the combination of anti-PD-1 and AV-MEL-1.

DETAILED DESCRIPTION:
The sequence is as follows:

1. Patients will provide consent for collection of blood and tumor, willingness to undergo leukapheresis, and intended plan to treat with a standard anti-PD-1 monotherapy regimen, and to treat with their patient-specific AV-MEL-1 once it has been manufactured.
2. Prior to starting anti-PD-1 therapy

   1. Surgically resected tumor tissue will be sent to AIVITA Biomedical where it will be processed to establish a short-term cell line of autologous tumor cells. Approximately 1 cm3 of surgically excised tumor is preferred. Whenever possible the tissue should be obtained from a lesion no greater than 2 cm in longest diameter. Part of the sample should be assessed by pathologists to confirm melanoma and to test for PDL-1 expression.
   2. Patients will undergo leukapheresis to obtain PBMC that will be converted into dendritic cells (DC).
   3. Patients who did not have a PET/CT or CT scan performed within the previous 6 weeks, will undergo a PET/CT or CT to define baseline disease status (measurable disease, non-measurable detectable disease, or no evidence of disease).
3. Patients will initiate anti-PD-1 therapy monotherapy (e.g. pembrolizumab or nivolumab) using standard doses and schedules of administration at week 0.
4. When the vaccine is ready, (approximately week 8 or 9) and the patient has had the opportunity to have received about two months of anti-PD-1 monotherapy,

   1. The patient will undergo radiographic assessment (PET/CT or CT) to classify disease status (measurable disease, non-measurable detectable disease, or no evidence of disease) and response (if there was measurable disease at baseline) to the anti-PD-1 therapy.
   2. AV-MEL-1 will be given concurrently with continuation of the anti-PD-1 therapy. AV-MEL-1 injections will be given weekly for 3 weeks, (weeks 10-12, then monthly at weeks 16, 20, 24, 28, and 32). Blood will be collected from patients prior to each injection for immune monitoring tests. The timing of AV-MEL-1 injections is not synchronized with the administration of anti-PD-1, but they can be administered on the same day.
5. If anti-PD-1 therapy is discontinued during vaccine treatment, the remaining vaccine doses may still be administered at the discretion of the patient's managing physician.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Karnofsky Performance Status (KPS) of > 70
* Presence of at least one metastatic lesion that is to be removed surgically as part of standard care (e.g. diagnosis or diagnostic testing, mono- or oligometastatic disease, alleviation of symptoms etc)
* • Diagnosis of metastatic melanoma with at least one lesion that is amenable for surgical resection per standard of care (e.g. diagnosis or diagnostic testing, mono- or oligometastatic disease, alleviation of symptoms etc)
* Considered appropriate for standard anti-PD1 antibody monotherapy by managing physician
* Given written informed consent to participate in the study

Exclusion Criteria:

* Known to have active hepatitis B or C or HIV (need not be screened)
* KPS of < 70; see Appendix A
* Known underlying cardiac disease associated with myocardial dysfunction that requires active medical treatment, or unstable angina related to atherosclerotic cardiovascular disease, or under treatment for arterial or venous peripheral vascular disease
* Diagnosis of any other invasive cancer or other disease process which is considered to be life-threatening within the next five years, and/or taking anti-cancer therapy for cancer other than melanoma
* Active infection that could be eminently life-threatening or other active medical condition that could be eminently life-threatening, including active blood clotting or bleeding diathesis.
* Known autoimmune disease, immunodeficiency, or disease process that involves the chronic or intermittent use of immunosuppressive therapy
* Uncontrolled brain or spinal cord metastases or active leptomingeal metastatic disease.
* Received another investigational drug within 28 days of the first dose or are planning to receive another investigational drug while receiving this investigational treatment
* Known hypersensitivity to GM-CSF
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Number of grade 3-5 adverse events with AV-MEL-1 + PD-1 versus PD-1 alone | 3 years
  Determine whether combining AV-MEL-1 with anti-PD-1 is associated with increased risk as defined by AEs per NCI common toxicity criteria

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Dillman, MD, Study Chair — Aivita Biomedical, Inc.
Locations (2):
- United States (2):
  - Jericho Rabago, Irvine, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California